CLINICAL TRIAL: NCT00745888
Title: Oxidative Stress in Critical Ill Patients in Surgical Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yu-Chang Yeh, National Taiwan University Hospital
Other Study IDs: 9561709132
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-08

CONDITIONS: Sepsis; Shock
Keywords: oxidative stress; intensive care; Postoperative intensive care
MeSH Terms: conditions — Sepsis; Shock

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: age > 18 y/o Patients admitted to surgical ICU
  Interventions: Other: Chemiluminescence Analyzer

INTERVENTIONS:
Other: Chemiluminescence Analyzer — measure reactive oxygen species

SUMMARY:
In clinical practice, the oxidative stress is related to circulatory shock, sepsis, acute lung injury, and acute respiratory distress syndrome. There are some questions on the oxidative stress of the critical illness. First, the investigators want to search out the effects of the past history, smoking, alcohol drinking, use of antioxidants, different diseases, and different duration of SIRS on the degree of oxidative stress. Second, besides total count of ROS, the investigators used new techniques to determine superoxide(O2●-), hydrogen peroxide (H2O2), and hypochlorous acid(HOCl). Furthermore, we want to investigate the correlation of the degree of different reactive oxygen species and the severity of SIRS or shock. Third, we try to investigate the correlation between the change of oxidative stress and the prognosis of the patients.

The investigators wish this study will help them to investigate the effect of oxidative stress on critical ill patients, to modulate the oxidative stress, to decrease the occurrence of SIRS, shock, and multiorgan failure, and to improve the long term outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y/o
* Admitted to surgical ICU

Exclusion Criteria:

* Patients with brain death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to surgical ICU
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
28-day Survival | 28 days

SECONDARY OUTCOMES:
Days stay in ICU Days on ventilator SOFA score Complications | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan